CLINICAL TRIAL: NCT04548479
Title: A Comparative Study of Incentive Spirometry and Positive Expiratory Pressure in Patients With Chest Trauma: a Randomized Controlled Trial
Brief Title: A Comparative Study of Incentive Spirometry and Positive Expiratory Pressure in Chest Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Granollers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Incentive Spirometry vs PEP
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Trauma Chest
MeSH Terms: conditions — Thoracic Injuries

STUDY DESIGN:
Intervention Model Description: aleatorizado 1:1
Who Masked: Outcomes Assessor
Masking Description: Los evaluadores de los resultados y el investigador que realiza la aleatorización
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEP group (Active Comparator): Chest physiotherapy depending on the location of the ribs fractures techniques are performed: 1. Postural control techniques; 2. Airways clearance techniques; 3. Breathing exercise (diaphragmatic breathing). 4. Early mobilization. 5. Positive expiratory pressure (PEP) breathing
  Interventions: Device: PEP bottle
- INS group (No Intervention): Chest physiotherapy depending on the location of the ribs fractures techniques are performed: 1. Postural control techniques; 2. Airways clearance techniques; 3. Breathing exercise (diaphragmatic breathing). 4. Early mobilization. 5. Inspiratory incentive spirometry breathing

INTERVENTIONS:
Device: PEP bottle — PEP bottle: it will be performed with a bottle of distilled water and a plastic tube, where the patient breathes against a resistance during expiration.
  Arms: PEP group

SUMMARY:
Chest trauma (CT) patients with 3 or more ribs fractures with or without pleuropulmonary injury are an indicator of severity. Chest physiotherapy (CP) and analgesia is the first line treatment in these patients.

The aim study is to evaluate the effect of positive expiratory pressure (PEP) breathing compared to the incentive spirometry in terms of pain control in the recent phase of CT.

DETAILED DESCRIPTION:
After acceptance to participate in the study, patients will be computerized randomized into 2 groups:

* PEP group: positive expiratory pressure (PEP) breathing.
* INS group: inspiratory incentive spirometry breathing. The period between day 0 and 20 days post-trauma is considered an immediate phase of TT.

Once admitted, an initial evaluation by the doctor will be performed, and pleuro-pulmonary complications, the presence of respiratory failure, and pain control will be evaluated. The CP will perform a clinical, pain control, secretion and a dynamic costal examination. The medical treatment of pain control will begin, and the treatment of CP will begin, where it will be randomized in 2 groups: 1- PEP group: positive expiratory pressure (PEP) breathing the help of a PEP bottle device. 2- INS group: inspiratory incentive spirometry device (Coach®). Will be daily FR sessions, on weekdays. Upon admission, hospital discharge and post-discharge, radiological checks (simple radiography) will be performed and forced vital capacity will be measured with forced spirometry.

ELIGIBILITY:
Inclusion Criteria:

* Chest trauma of 3 or more rib fractures with or without hemopneumothorax
* Signed informed consent.

Exclusion Criteria:

* Non-collaborating patients.
* Failure to submit a duly completed follow-up sheet for carrying out a minimum daily guideline (3 times a day) for CP treatment.
* Presence of respiratory failure at admission: PaO2 <60mmHg and / or PaCO2> 50mmHg.
* Medical indication for invasive or non-invasive ventilatory support.
* Presence of undrained pneumothorax.
* Complications that limit early mobility.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Improve the degree of pain | 1 month
  To assess if PEP decreased pain

SECONDARY OUTCOMES:
Resolution of pleural lesions | 1 month
  To analysed if PEP allows faster resolution of pleural lesions
Improve lung function | 1 month
  To determined if PEP improves functional sequelae secondary to thoracic trauma.
Reduce hospital stay | 1 month
  To assess if PEP decreased hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Gemma Molist, Study Chair — Hospital de Granollers
Locations (1):
- Inmaculada Castillo, Seva, Barcelona, Spain

REFERENCES:
- [Background] Overend TJ, Anderson CM, Lucy SD, Bhatia C, Jonsson BI, Timmermans C. The effect of incentive spirometry on postoperative pulmonary complications: a systematic review. Chest. 2001 Sep;120(3):971-8. doi: 10.1378/chest.120.3.971. PMID 11555536
- [Background] Simon B, Ebert J, Bokhari F, Capella J, Emhoff T, Hayward T 3rd, Rodriguez A, Smith L; Eastern Association for the Surgery of Trauma. Management of pulmonary contusion and flail chest: an Eastern Association for the Surgery of Trauma practice management guideline. J Trauma Acute Care Surg. 2012 Nov;73(5 Suppl 4):S351-61. doi: 10.1097/TA.0b013e31827019fd. PMID 23114493
- [Background] Unsworth A, Curtis K, Asha SE. Treatments for blunt chest trauma and their impact on patient outcomes and health service delivery. Scand J Trauma Resusc Emerg Med. 2015 Feb 8;23:17. doi: 10.1186/s13049-015-0091-5. PMID 25887859
- [Background] Gunduz M, Unlugenc H, Ozalevli M, Inanoglu K, Akman H. A comparative study of continuous positive airway pressure (CPAP) and intermittent positive pressure ventilation (IPPV) in patients with flail chest. Emerg Med J. 2005 May;22(5):325-9. doi: 10.1136/emj.2004.019786. PMID 15843697
- [Background] Sehlin M, Ohberg F, Johansson G, Winso O. Physiological responses to positive expiratory pressure breathing: a comparison of the PEP bottle and the PEP mask. Respir Care. 2007 Aug;52(8):1000-5. PMID 17650355